CLINICAL TRIAL: NCT03567356
Title: Medication Adherence Therapy - Psychosocial Leverage Using a Treatment Significant Other
Brief Title: Treatment of Opioid Use: Medication Adherence Therapy
Acronym: MAT-PLUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Potomac Health Foundations (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MTC002
Record Dates: First submitted 2018-05-31; First posted 2018-06-25 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Opioid Dependence; Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Open-label Treatment as Usual vs. Intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment as Usual (No Intervention): TAU will contain patients who will be receiving treatment for opioid use disorder through their usual venues without the family engagement, assertive outreach, and home delivery of XRNTX doses.
- MAT-Plus Intervention (Experimental): The intervention group will receive the multi-component MAT-PLUS treatment: 1) Significant other engagement through the "Helping Hands" approach empowers designated concerned helpers, providing concrete guidance for monitoring, supervision, and improving adherence for their loved one in treatment; 2) Care coordination and case management by counselors to enhance adherence to XRNTX ; 3) Assertive outreach incorporates frequent multi-channel outreach with the goal of achieving XRNTX dosing.
  Interventions: Other: MAT-PLUS "Helping Hands"

INTERVENTIONS:
Other: MAT-PLUS "Helping Hands" — 1) Significant other engagement through the "Helping Hands" approach empowers designated concerned helpers, providing concrete guidance for monitoring, supervision, and improving adherence for their loved one in treatment; 2) Care coordination and case management by counselors to enhance adherence to XRNTX ; 3) Assertive outreach incorporates frequent multi-channel outreach with the goal of achieving XRNTX dosing.
  Arms: MAT-Plus Intervention

SUMMARY:
To test the feasibility and acceptability of a novel approach for improving the delivery and effectiveness of XRNTX treatment for opioid use disorder (OUD) - the MAT-PLUS intervention. The components of the MAT-PLUS intervention are: XRNTX, initiated during an episode of inpatient/residential treatment and dosed monthly, provides opioid receptor blockade, relapse prevention and overdose prevention; Significant other engagement empowers family members or other designated concerned others, providing concrete guidance for monitoring, supervision, and improving adherence for their loved one in treatment; Assertive outreach incorporates frequent multi-channel outreach, in a model that specifically targets engagement and motivation for medication adherence; Counselor care coordination and case management focused on medication management and adherence. This objective #1 will be accomplished by conducting a small-scale, 2-arm, open label, RCT pilot study of 4 months of treatment with the MAT-PLUS intervention (significant other engagement and training, medication care coordination by counselors, assertive outreach) + TAU (monthly doses of XRNTX + routine counseling), vs TAU for n=40 (20 per arm) patients with OUD. Adult patients ages 18+ who receive an initial dose of XRNTX during an index episode of inpatient/residential/detox treatment for opioid addiction at a public-sector community treatment program treatment, with intention to continue in outpatient treatment. The experimental arm will receive the MAT-PLUS intervention for 4 months of ongoing outpatient treatment with XRNTX. The control arm will receive 4 months of standard TAU (XRNTX + clinic-based counseling) without MAT-PLUS. At the beginning of the trial an additional small (N = 4 or 5) group of test patients will receive the MAT-PLUS intervention to test and refine the study procedures.

DETAILED DESCRIPTION:
Residential detox is an ideal opportunity for initiation of relapse prevention medication, particularly XRNTX, which requires some delay after recent opioid use. But concerns from the field emphasize barriers to induction (as highlighted by the recent results of the CTN51 XBOT study), poor adherence and retention. Clarification is needed on optimal delivery, including a psychosocial treatment platform that is focused more specifically on medication adherence through engagement and empowerment of significant others, and through training and supervision of counselors. Adherence in non-research conditions has been a barrier. To address these gaps, it is proposed this robust intervention, incorporating XRNTX into a multi-component model of care emphasizing adherence enhancement. Assertive outreach is a well-described intervention that is effective in chronic illness, eg in the Assertive Community Treatment (ACT) model for serious and persistent mental illness, and the Integrated Dual Disorder Treatment (IDDT) model for co-occurring disorders. Significant other involvement is a well-established method of improving adherence (e.g. in Network Therapy and Community Reinforcement Approach and Family Training). Significant other involvement is also built into the standard Medication Management model (used in XBOT,COMBINE and others) but it has not been actually used in most implementations. Finally, the use of counselors to drive medication adherence takes advantage of the typically greater contact and alliance that counselors have with patients compared to medical staff.

Several adherence enhancement components are combined synergistically: XRNTX, initiated during residential treatment and dosed monthly; significant other engagement empowers caregivers, providing guidance for encouragement, monitoring and supervision of medication adherence; Assertive outreach incorporates frequent multi-channel contact, case management; Counselor role clarification, training and supervision provides a clear focus on medication adherence.

Primary outcome for this objective is # of doses of XRNTX received within the planned 4 months duration of outpatient treatment. The primary analysis will be a comparison of the mean # of doses in the intervention compared to the control group. Additional analyses will include comparisons of % of subjects receiving all 4 doses, % of subjects receiving at least 1 dose as outpatients as a demonstration of linkage from inpatient to outpatient treatment.

Secondary outcomes for this feasibility objective include process outcomes for feasibility and acceptability, including: # and type of outreach attempts (phone call, email, text, facebook message, etc) and successful contacts with patients and significant others, utilization of TAU counseling, rates of return to treatment after dropout. Lastly, assessments of satisfaction and significant other involvement will be obtained through focus groups conducted separately with patients and significant others to assess qualitative acceptability factors, both barriers and facilitators to success.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18+ with OUD who present for an index episode of residential/inpatient opioid detoxification and seek treatment with XRNTX at community treatment provider Mountain Manor Treatment Center (MMTC)

Exclusion Criteria:

* LFTs > 5x ULN
* Psychiatric or medical instability (eg suicidality, psychosis. Sickle Cell disease with frequent crises, etc) that would preclude participation in the trial
* Living situation (location greater than 60 miles from the center, homelessness) that that would preclude participation in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Mean number of XRNTX doses within each group | 4 months
  Mean Number of XRNTX doses received within 4 months of study

SECONDARY OUTCOMES:
Rate of opioid relapse during the study period | Data measured every 2 weeks for the duration of the study period
  Relapse = 10 days of use within a 28 day period. Days of opioid use will be assessed through urine toxicology and self report methods.
Percent Linkage to continuing care | 1 month
  Percent receiving initial outpatient dose
Mean Number of days of opioid use | 4 months
  Mean number of opiate using days in each group

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fishman, MD, Principal Investigator — Maryland Treatment Centers/PHF
Locations (1):
- Mountain Manor Treatment Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wenzel K, Thomas J, Carrano J, Stidham J, Fishman M. A pilot randomized controlled trial of medication adherence therapy: Psychosocial leverage using a significant other (MAT-PLUS) for individuals on extended-release naltrexone. J Subst Use Addict Treat. 2024 Aug;163:209366. doi: 10.1016/j.josat.2024.209366. Epub 2024 Apr 16. PMID 38636807